CLINICAL TRIAL: NCT01952704
Title: A Randomized Controlled Trial of Aerobic Exercise to Improve Memory in TBI
Brief Title: Aerobic Exercise to Improve Memory in TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Brain Injury Research (Other)
Responsible Party: Principal Investigator, Victoria Leavitt, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-687-11
Record Dates: First submitted 2013-09-24; First posted 2013-09-30 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise (Experimental): 30 minutes x 3 times/week x 12 weeks of stationery cycling
  Interventions: Behavioral: Aerobic exercise
- Non-aerobic exercise (Placebo Comparator): 30 minutes x 3 times/week x 12 weeks of gentle non-aerobic stretching
  Interventions: Behavioral: Placebo control

INTERVENTIONS:
Behavioral: Aerobic exercise
  Arms: Aerobic exercise
Behavioral: Placebo control — Non-aerobic stretching sessions will be conducted 3x/week for 30 minutes over 12 weeks.
  Arms: Non-aerobic exercise

SUMMARY:
Aerobic exercise holds a multitude of health benefits. Studies in mice have shown that aerobic exercise improves memory, and increases the volume of the hippocampus, the brain's primary memory center. Only two studies have been conducted in humans, one in healthy elders, and the other in a schizophrenia population. So far, there has never been an aerobic exercise trial in traumatic brain injury (TBI) to look at hippocampal volume and memory as outcomes of interest. The proposed project is a randomized controlled trial of aerobic exercise in persons with TBI. We will conduct a 12-week (36 sessions) program of aerobic exercise (stationary cycling), versus a control condition of non-aerobic exercise (stretching), in memory-impaired TBI patients to a) increase hippocampal volume and b) improve memory. Importantly, we also expect benefits of aerobic exercise on the level of brain function. Specifically, we will look at 'functional connectivity,' which refers to how efficiently remote regions of the brain 'talk' to each other. TBI is an ideal population to benefit from aerobic exercise, given the young age at which many individuals sustain TBI, which allows for benefits of aerobic exercise to be maximally realized in a population with sufficient neurofunctional reserve. The expected benefits of aerobic exercise (increased hippocampal volume, improved memory) from this intervention stand to have a meaningful impact on people with TBI, including improved health, productivity, independence, and quality of life. And, unlike current treatments for memory impairment (e.g., pharmacological agents, cognitive rehabilitation), aerobic exercise is a cost-effective, all natural, readily-available treatment for memory problems.

ELIGIBILITY:
Inclusion Criteria:

* TBI greater than or equal to 1 year
* MRI compatibility
* Right Handed

Exclusion Criteria:

* Reported lower body weakness or use of an assistive device for walking
* History of pulmonary disease, heart disease, vascular disease of the legs, high blood pressure
* History of stroke, other neurological disease/disorder, serious psychiatric illness
* Engaging in more than 30 minutes of aerobic exercise per week
* Current use of steroids, benzodiazepines, and/or neuroleptics
* History of substance abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Hippocampal volume | 1 week post intervention
  Volumetric software will be used to measure hippocampus at baseline and follow-up (within 1 week of completion of 12-week intervention).